CLINICAL TRIAL: NCT01241071
Title: Effects of a Myofascial Release Protocol on Pain, Disability and Activation Pattern of Erector Spinae in Patients With Chronic Low Back Pain
Brief Title: Effects of Myofascial Release on Pain, Disability and Electromyography of Erector Spinae in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: Hospital Arnau de Vilanova (Other)
Responsible Party: Principal Investigator, Eva Segura Ortí, PhD, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEU-UCH-88
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Low Back Pain; Disability; Motor Activity; Range of Motion
Keywords: Lumbar region; Pain; Fascia; Electromyography; Goniometry
MeSH Terms: conditions — Low Back Pain; Motor Activity; Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Myofascial treatment (Experimental): Myofascial release techniques of different muscles implicated in low back pain
  Interventions: Other: myofascial treatment
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: myofascial treatment — myofascial release techniques of different muscles implicated in low back pain
  Arms: Myofascial treatment
Other: Placebo — A manual sham intervention will be applied to different muscles implicated in low back pain
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether myofascial release techniques are effective in the improvement of pain, disability and electromyography response of lumbar muscles in patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* low back pain for more than 3 months

Exclusion Criteria:

* vertebra fractures
* systemic disease (spondylitis, neoplasia, infectious, vascular, endocrine or metabolic disorders)
* spinal surgery
* advanced lumbar instability
* osteoporosis (in advanced stage)
* degenerative articular disease
* acute soft tissue inflammation
* rheumatoid arthritis
* osteomyelitis
* neuromuscular disease
* lower limb musculoskeletal injuries
* radiculopathy
* cauda equine syndrome
* myelopathy
* stenosis
* structural spine deformity (kyphoscoliosis...)
* pregnancy
* abundant menstruation
* IUD carrier
* mental disease
* dermatologic disease
* skin sensitivity
* aneurysma
* corticosteroids treatment
* anticoagulant therapy
* hypertension
* diabetes
* hemophilia
* leucemia
* rejection to manual contact

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Lumbar Pain | 3 weeks
  Short Form McGill Pain Questionnaire. Visual Analogical Scale

SECONDARY OUTCOMES:
Disability | 3 weeks
  Roland Morris Disability Questionnaire
Fear Avoidance Beliefs | 3 weeks
  Fear Avoidance Beliefs Questionnaire
EMG Erector Spinae | 3 weeks
  Electromyography record (MEGAWIN 6000)
Lumbar ROM | 3 weeks
  Electrogonyometry Fastrak (Polhemus)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Romero, Dean, Study Director — Health Science Faculty CEU-UCH
Locations (1):
- CEU Cardenal Herrera University, Moncada, Valencia, Spain

REFERENCES:
- [Background] FLOYD WF, SILVER PH. Function of erectores spinae in flexion of the trunk. Lancet. 1951 Jan 20;1(6647):133-4. doi: 10.1016/s0140-6736(51)91212-3. No abstract available. PMID 14795792
- [Background] Alschuler KN, Neblett R, Wiggert E, Haig AJ, Geisser ME. Flexion-relaxation and clinical features associated with chronic low back pain: A comparison of different methods of quantifying flexion-relaxation. Clin J Pain. 2009 Nov-Dec;25(9):760-6. doi: 10.1097/AJP.0b013e3181b56db6. PMID 19851155
- [Background] Grinnell F. Fibroblast mechanics in three-dimensional collagen matrices. J Bodyw Mov Ther. 2008 Jul;12(3):191-3. doi: 10.1016/j.jbmt.2008.03.005. Epub 2008 May 23. PMID 19083673
- [Background] Fernandez-Perez AM, Peralta-Ramirez MI, Pilat A, Villaverde C. Effects of myofascial induction techniques on physiologic and psychologic parameters: a randomized controlled trial. J Altern Complement Med. 2008 Sep;14(7):807-11. doi: 10.1089/acm.2008.0117. PMID 18724827
- [Background] Schleip R, Klingler W, Lehmann-Horn F. Active fascial contractility: Fascia may be able to contract in a smooth muscle-like manner and thereby influence musculoskeletal dynamics. Med Hypotheses. 2005;65(2):273-7. doi: 10.1016/j.mehy.2005.03.005. PMID 15922099
- [Background] Saiz-Llamosas JR, Fernandez-Perez AM, Fajardo-Rodriguez MF, Pilat A, Valenza-Demet G, Fernandez-de-Las-Penas C. Changes in neck mobility and pressure pain threshold levels following a cervical myofascial induction technique in pain-free healthy subjects. J Manipulative Physiol Ther. 2009 Jun;32(5):352-7. doi: 10.1016/j.jmpt.2009.04.009. PMID 19539117
- [Background] Ritvanen T, Zaproudina N, Nissen M, Leinonen V, Hanninen O. Dynamic surface electromyographic responses in chronic low back pain treated by traditional bone setting and conventional physical therapy. J Manipulative Physiol Ther. 2007 Jan;30(1):31-7. doi: 10.1016/j.jmpt.2006.11.010. PMID 17224353
- See also: CEU Cardenal Herrera University is the first private university in the Valencian Community. It belongs to the San Pablo CEU Foundation which is a leading educational organization in Spain with three universities all over Spain. — http://www.uchceu.es